CLINICAL TRIAL: NCT06488274
Title: Assessment of the Evolution of functIonal Gastrointestinal Disorders in Infants During Their Dietary Management With a New Infant Formula
Brief Title: Evolution of Functional Gastrointestinal Disorders in Infants Fed With a New Infant Formula
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Collaborators: Axiodis CRO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UP2022_FGID
Record Dates: First submitted 2024-06-21; First posted 2024-07-05 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Regurgitations; Colic; Constipation; Infant formula; GIGER scale; Nutrition; Infants
MeSH Terms: conditions — Gastrointestinal Diseases; Gastroesophageal Reflux; Colic; Constipation

STUDY DESIGN:
Intervention Model Description: Interventional, open-label, non-comparative multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test formula (Experimental): The test product is a thickened infant formula containing symbiotic (fibers and probiotics)
  Interventions: Dietary Supplement: New infant formula

INTERVENTIONS:
Dietary Supplement: New infant formula — The new formula will be given to infants during the 4-month study period.

SUMMARY:
This study aims to assess the evolution of functional gastrointestinal disorders (FGIDs) in infants fed with a new infant formula, using the Gastrointestinal (GI) and gastroesophageal reflux (GER) (GIGER) scale through an interventional, open-label, non-comparative multicenter study.

DETAILED DESCRIPTION:
The study comprises a first period of 30 days followed by an optional intervention period of 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Infants presenting with at least one of the FGIDs below, defined based on adapted Rome IV criteria as follows:

   1.1 Regurgitations: 1.2 Colic: 1.3 Constipation:
2. Infants born at 35 weeks or more of gestational age
3. Infants up to 4 months of age

Exclusion Criteria:

1. Exclusively or partially breastfed infants (i.e. > 2 breast feeds per day) with maternal willingness to continue breastfeeding
2. Diversified infants or whose parents intend to start diversification within the first 2 weeks of the study
3. Use of antibiotics at inclusion visit (V0) and within 7 days before the inclusion visit (V0)
4. The willingness to take additional pre-, probiotics or thickening agents during the study
5. Known allergy/intolerance to any of the product ingredients or suspected allergy to cow's milk requiring an eviction diet
6. Infants presenting with any other situation including the participation in another clinical trial, which, according to the investigator, may interfere with the study participation, or lead to a particular risk for the patient

(non exhaustive list)

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 139 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the Gastrointestinal and Gastroesophageal Reflux (GIGER) scale score | Day 30
  The main outcome will be the evolution of the sum score of the Gastrointestinal and Gastroesophageal Reflux (GIGER) scale (Pados et al., 2021). The GIGER score varies from 0 to 180 being the worst.

SECONDARY OUTCOMES:
Evolution of FGIDs (regurgitations, colic and constipation) | Day 14, Day 30, Day 60, Day 90, Day 120
  FGIDs such as regurgitation, colic and constipation will be assessed according to adapted Rome IV criteria. The improvement and complete resolution timeframe of each FGID present at inclusion and/or occurring during the study will be determined.
Regurgitation frequency | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  The number of daily regurgitation episodes and the daily volume of regurgitation will be assessed on average over the last 3 days. The frequency of regurgitations away from meals and of continuous regurgitations of small volumes after feeding will be assessed on average over the last 3 days via a 4-point scale [Never; Rarely; Often; Always].
Regurgitation severity | Day 14, Day 30, Day 60, Day 90, Day 120
  The regurgitation severity will be assessed using the adapted Vandenplas regurgitation score (from 0 to 6 being the worst) (Vandenplas et al., 1994) over the last 3 days preceding each visit.
Stool frequency and consistency in non constipated infant | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  If the infant is not constipated at inclusion and during the study, the average main stool consistency will be assessed based on the BITSS scale (Brussels Infant and Toddler Stool Scale) as well as the daily average number of stools over the last 3 days.
  The BITTS scale is a reliable instrument to assess stools of non-toilet trained children. It consists of 7 color photographs of diapers containing stools from infants and toddlers categorized as Hard, Formed, Loose, or Watery (Huysentruyt et al., 2019).
Stool frequency and consistency in constipated infant | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  If the infant is constipated at one visit during the study, the total number of each stool consistency will be assessed for the next visit based on the BITSS scale over the last 7 days. The total number of stools over the last 7 days will be calculated.
Defecation pain frequency in constipated infant | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  If the infant is constipated at one visit during the study, the frequency of defecation pain will be assessed for the next visit based on a 3-point scale (No; Yes, only 1 time; Yes, >1 time) over the last 7 days.
Colic | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  Colic will be assessed through unexplained crying duration and fussing/irritability duration on average over the last 3 days and reported based on a 4-point scale (< 1h; 1h-2h; 2h-3h; > 3h).
Gas/flatulence severity | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  Gas/flatulence severity will be assessed on average over the last 3 days using a visual analog scale (from 0=No symptom to 10=Very severe symptoms).
Abdominal distension severity | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  Abdominal distension is defined as a swollen, tense and hard to the touch stomach. Its severity will be assessed on average over the last 3 days using a visual analog scale (from 0=No symptom to 10=Very severe symptoms).
GIGER score | Day 7, Day 14, Day 60, Day 90, Day 120
  Evolution of Gastrointestinal and Gastroesophageal Reflux (GIGER) scale total score (from 0 to 180) and 3 subscores (subscore 1: from 0 to 75; subscore 2: from 0 to 65; subscore 3: from 0 to 40) from baseline. The higher the GIGER is, the worst the symptoms are.
Investigator's evaluation of the evolution of FGIDs | Day 14, Day 30, Day 60, Day 90, Day 120
  The investigator will evaluate the evolution of each FGID (i.e. regurgitations, constipation, colic) using a 4-point scale (Improvement; Worsening; No evolution; Not applicable) over the past period.
Number of bottles at night | D7, D14, D30, D60, D90, D120
  The number of bottles at night will be recorded on average over the last 3 days.
Sleep | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  The average sleep duration will be reported over the last 3 days and sleep quality will be assessed using a visual analog scale (from 0= Difficult to fall asleep, frequent awakenings to 10= Easy and quick falling asleep, no awakenings without obvious cause).
Infant's quality of life | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  Parents will complete the QUALIN questionnaire (score from -68 to +68) (Manificat et al., 2000) over the last week.
Weight | Day 30, Day 60, Day 90, Day 120
  Weight will be expressed in kg and in z scores according to the World Health Organization (WHO) Child Growth Standards.
Height | Day 30, Day 60, Day 90, Day 120
  Height will be expressed in cm and in z scores according to the WHO Child Growth Standards.
Head circumference | Day 30, Day 60, Day 90, Day 120
  Head circumference will be expressed in cm and in z scores according to the WHO Child Growth Standards.
BMI | Day 30, Day 60, Day 90, Day 120
  BMI will be expressed in value and z scores according to the WHO Child Growth Standards.
Adverse events | Through study completion (up to 30 days or 120 days if participation to the optional intervention period)
  Any untoward medical reaction occuring from the signatture of the consent until the end of the participant's participation
Parents' satisfaction | Day 7, Day 14, Day 30, Day 60, Day 90, Day 120
  Parents' satisfaction will be assessed on the product use and acceptability using a 5-point Likert scale and more specifically on the evolution of each FGID (i.e. regurgitations, constipation, colic) using a 4-point scale (Improvement; Worsening; No evolution; Not applicable) over the past period.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Batard, Dr., Study Director — Ambulatory pediatrician in Vincennes (France); Camille Jung, Prof., Study Chair — Centre Hospitalier Intercommunal (CHI) in Créteil (France)
Locations (4):
- France (4):
  - Site 02, Nice
  - Site 04, Paris
  - Site 03, Toulon
  - Site 01, Vincennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pados BF, Repsha C, Hill RR. The Gastrointestinal and Gastroesophageal Reflux (GIGER) Scale for Infants and Toddlers. Glob Pediatr Health. 2021 Jul 14;8:2333794X211033130. doi: 10.1177/2333794X211033130. eCollection 2021. PMID 34350308
- [Background] Vandenplas Y, Hachimi-Idrissi S, Casteels A, Mahler T, Loeb H. A clinical trial with an "anti-regurgitation" formula. Eur J Pediatr. 1994 Jun;153(6):419-23. doi: 10.1007/BF01983405. PMID 8088297
- [Background] Huysentruyt K, Koppen I, Benninga M, Cattaert T, Cheng J, De Geyter C, Faure C, Gottrand F, Hegar B, Hojsak I, Miqdady M, Osatakul S, Ribes-Koninckx C, Salvatore S, Saps M, Shamir R, Staiano A, Szajewska H, Vieira M, Vandenplas Y; BITSS working group. The Brussels Infant and Toddler Stool Scale: A Study on Interobserver Reliability. J Pediatr Gastroenterol Nutr. 2019 Feb;68(2):207-213. doi: 10.1097/MPG.0000000000002153. PMID 30672767
- [Background] Manificat S, Dazord A, Langue J, Danjou G, Bauche P, Bovet F, Cubells J, Luchelli R, Tockert E, Conway K. [Evaluation of the quality of life of infants and very young children: validation of a questionnaire. Multicenter European study]. Arch Pediatr. 2000 Jun;7(6):605-14. doi: 10.1016/s0929-693x(00)80127-x. French. PMID 10911526